CLINICAL TRIAL: NCT01937598
Title: Antidiabetic Effects of Adding a DPP-4 Inhibitor (Sitagliptin) to Pre-Existing Treatment With an Incretin Mimetic (Liraglutide) in Patients With Type 2 Diabetes Treated With Metformin
Brief Title: Antidiabetic Effects of Adding a DPP-4 Inhibitor to Pre-Existing Treatment With an Incretin Mimetic in Patients With T2D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Michael A. Nauck (Other)
Responsible Party: Sponsor-Investigator, Michael A. Nauck, Prof. Dr. med., Diabeteszentrum Bad Lauterberg im Harz
Organization: Diabeteszentrum Bad Lauterberg im Harz (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 120-0569-DZBL-2012; 2013-001764-35 (EudraCT Number)
Record Dates: First submitted 2013-08-27; First posted 2013-09-09 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes
Keywords: Incretin, DPP-4 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin, then Placebo (Experimental)
  Interventions: Drug: Placebo; Other: Mixed meal test; Drug: Liraglutide; Drug: Sitagliptin
- Placebo, then Sitagliptin (Experimental)
  Interventions: Drug: Placebo; Other: Mixed meal test; Drug: Liraglutide; Drug: Sitagliptin

INTERVENTIONS:
Drug: Placebo — Patients administered a single dose of placebo during a mixed meal challenge.
Other: Mixed meal test — Subjects will be instructed to consume the mixed meal test within 20 minutes. The exact start and stop time of the mixed meal test consumption will be recorded in the CRF. The mixed meal test procedures will be identical for all subjects randomised in the study. To detect the plasma glucose excursion after mixed meal test, plasma glucose will be closely monitored
Drug: Liraglutide — Patients on metformin monotherapy will, after screening and randomization, enter a run-in period of 2 weeks with the additional treatment of liraglutide (0.6 mg/d for 1 week followed by 1.2 mg/d for another week) that will be continued for the entire duration of the study.
  Other Names: Victoza
Drug: Sitagliptin — Patients administered a single dose of Sitagliptin during a mixed meal challenge.

SUMMARY:
Objectives: To quantify differences in control of glycemia (primary objective) and the secretion of endogenous incretin hormones (secondary objective) comparing sitagliptin or placebo added to pre-existing therapy with liraglutide and metformin

DETAILED DESCRIPTION:
This is a double blind, controlled, cross-over comparison of adding sitagliptin (or placebo) to pre-existing metformin+liraglutide therapy. Patients with type 2 diabetes mellitus (T2DM) on pre-existing treatment with metformin (≥ 1500 mg/d) monotherapy or metformin plus liraglutide (1.2 mg/d) will be studied. Patients on metformin monotherapy will, after screening and randomization, enter a run-in period of 2 weeks with the additional treatment of liraglutide (0.6 mg/d for 1 week followed by 1.2 mg/d for another week). At the end of this 2 weeks therapy, a mixed meal challenge will take place, with the assessment of glucose and hormone responses (insulin, C-peptide, glucagon, GLP-1 [glucagon-like peptide-1], GIP (gastric inhibitory peptide) and gastric emptying as measured by 13C (carbon 13)-octanoate breath tests. Prior to the meal tests, liraglutide will be administered at a dose of 1.2 mg per injection, which is the recommended dose for treatment. Sitagliptin will be used at a dose of 100 mg, which is recommended for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Signed & dated written informed consent
* Male & female subjects with a diagnosis of type 2 diabetes mellitus according to ADA criteria at least 4 months prior to screening
* Medical history without major pathology (with the exception of type 2 diabetes) as judged by the investigator
* On a stable regimen of metformin for at least 1 month and liraglutide 1.2 mg for at least 1 week at the time-point of randomisation.
* Age: 25 - 75 years, both inclusive
* Body mass index (BMI): 22 - 40kg/m^2, both inclusive
* HbA1c ≥ 6.5 and ≤ 8.5% (≥ 7.0 and ≤ 8.5% for patients without previous liraglutide treatment)
* Female must be post-menopausal, surgically sterilized or practicing an effective birth control

Exclusion criteria

* Subjects with type 1 diabetes, maturity onset diabetes of the young (MODY) or secondary forms of diabetes such as due to pancreatitis
* Current or previous treatment with insulin therapy (except for treatment at diabetes' diagnosis, within a clinical trial, for surgical procedures or during an acute illness, and no insulin administration within the 6 months before screening)
* Treatment with any hypoglycaemic medication other than metformin and liraglutide within one month prior to screening
* Known of diabetic gastroparesis and / or prokinetic therapy
* Subjects that underwent surgery of the upper gastrointestinal tract
* Women who are pregnant, intending to become pregnant during the study period, currently lactating females, or women of child-bearing potential not using highly effective, medically approved birth control methods
* Any severe medical or surgical history of conditions likely to confound study assessments or study endpoints, for example but not limited to haemoglobinopathies, inflammatory bowel disease, cystic fibrosis, bariatric surgery and/or any surgery shortening the intestine, history of lactose intolerance, lactose- or glucose-galactose-malabsorption
* A suspicion of medullary thyroid cancer or a multiple endocrine neoplasia
* A personal or family history of medullar thyroid cancer or a multiple endocrine neoplasia
* Serious and/or unstable coronary heart disease (unstable angina, myocardial infarction within the preceding 6 months), congestive heart failure of New York Heart Association Class III or worse (severe limitation of physical activity; physical activity of low intensity resulting in fatigue, palpitation, or dyspnoea), second/third degree heart block, superior vena cava syndrome, uncontrolled hypertension, history of congenital QT-syndrome within family, history of stroke (within the preceding 6 months) or serious peripheral vascular disease
* History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (grade 3), left bundle branch block, or asymptomatic sustained ventricular tachycardia are not allowed
* Marked diabetic complications: severe autonomic or sensory neuropathy including previously diagnosed gastroparesis; proliferative retinopathy
* Any respiratory disease leading to respiratory insufficiency and/or depression including but not limited to clinically significant: bronchial asthma, chronic obstructive pulmonary disease, that might impact to the breath test, as judged by the investigator
* Clinically significant vital signs including known bradycardia with pulse rate < 50/min or 12-lead ECG findings including QTc (corrected QT interval) > 450 msec for males or QTc > 470 msec for women
* Clinically significant abnormal haematology, biochemistry, lipids, or urinalysis or coagulation screening tests, as judged by the Investigator
* Moderate or severe renal dysfunction defined as an estimated creatinine clearance (MDRD equation) GFR (glomerular filtration rate) <50 ml/min.
* Clinical or laboratory evidence of hepatic dysfunction or disease; laboratory evidence defined as any of the following parameters: alkaline phosphatase, ALT , AST or bilirubin > 3x ULN (upper Limit of normal). Isolated mild rise in bilirubin considered to be due to Gilbert's condition is allowed
* Uncontrolled high blood pressure (DBP (diastolic blood pressure) > 95 mmHg and/or SBP (systolic blood pressure) > 160 mmHg), unless clearly documented to be white-coat hypertension
* History of any psychiatric condition that might impair the subject's ability to understand or to comply with the requirements of the study or to provide informed consent
* History of relevant drug and/or food allergies or a history of severe anaphylactic reaction
* Currently active or history of alcohol abuse (defined as an intake of more than 24 units of alcohol per week; one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits) or drug addiction (including soft drugs like cannabis products)
* Use of concomitant medication which would be likely to interact with metformin, sitagliptin or liraglutide (according to the subject information leaflet). Participation in another study within the 3 months preceding screening or 5-half-lives of drug studied, whichever is longer, prior to study drug administration
* Malignancy within 5 years of study start, except for successfully treated local basal cell carcinomas
* Known to be positive for Hepatitis B surface antigen or Hepatitis C antibodies (or diagnosed with active hepatitis according to local practice)
* Subject who has donated or lost > 500 mL blood within 3 months prior to screening & has a Hb < 14 g/dl at screening
* History of hypersensitivity to the study drug or any of the excipients or to medicinal products with similar chemical structures
* Veins unsuitable for repeated venipuncture

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof. Dr., Principal Investigator — Diabeteszentrum Bad Lauterberg
Locations (1):
- Diabeteszentrum Bad Lauterberg, Bad Lauterberg im Harz, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin, Then Placebo: Participants first received Sitagliptin tablet before mixed meal test, after washout they then received Placebo before the mixed meal test.
- Placebo, Than Sitagliptin: Participants first received Placebo tablet before mixed meal test, after washout they then received Sitagliptin before the mixed meal test.
Period: Overall Study
Arm/Group | Sitagliptin, Then Placebo | Placebo, Than Sitagliptin
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants (cross-over design) received all interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11)
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Incremental Area Under the Plasma Glucose (BG) Concentration-time Profile (AUC)
Description: Incremental area under the plasma glucose (BG) concentration-time profile (AUC) immediately before to 300 min after a mixed meal test. In addition, the time course of BG values will be analysed with an ANCOVA model for repeated measurements with placebo baseline values as covariate. Time points to create the curce were 0, 15, 30, 45, 60, 90, 120, 150, 180, 240 and 300 minutes post mixed meal test.
Time Frame: 0 to 300 min post mixed meal test
Measure: Mean (Standard Error); unit: [mg*min/dL]
Groups:
- Sitagliptin: Substance: Sitagliptin phosphate H2O Pharmaceutical form: tablets Source: MSD SHARP & DOHME GMBH, Doses: 100 mg, Route of administration: p.o. as a tablet
  Sitagliptin
  Mixed meal test: Subjects will be instructed to consume the mixed meal test within 20 minutes. The exact start and stop time of the mixed meal test consumption will be recorded in the CRF(case report form). The mixed meal test procedures will be identical for all subjects randomised in the study. To detect the plasma glucose excursion after mixed meal test, plasma glucose will be closely monitored
  Liraglutide: Patients on metformin monotherapy will, after screening and randomization, enter a run-in period of 2 weeks with the additional treatment of liraglutide (0.6 mg/d for 1 week followed by 1.2 mg/d for another week) that will be continued for the entire duration of the study.
- Placebo: Substance: Placebo (sitagliptin) Pharmaceutical form: tablets Source: MSD SHARP & DOHME GMBH Doses: - Route of administration: p.o. as tablets
  Placebo
  Mixed meal test: Subjects will be instructed to consume the mixed meal test within 20 minutes. The exact start and stop time of the mixed meal test consumption will be recorded in the CRF. The mixed meal test procedures will be identical for all subjects randomised in the study. To detect the plasma glucose excursion after mixed meal test, plasma glucose will be closely monitored
  Liraglutide: Patients on metformin monotherapy will, after screening and randomization, enter a run-in period of 2 weeks with the additional treatment of liraglutide (0.6 mg/d for 1 week followed by 1.2 mg/d for another week) that will be continued for the entire duration of the study.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
[mg*min/dL] | 5678 (329) | 5557 (547)

2. Secondary Outcome: AUC Plasma Glucose
Description: Incremental AUC from 0 to 300 min
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: mmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
mmol/l*min | 315.4 (18.3) | 308.7 (30.4)

3. Secondary Outcome: AUC Insulin
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: nmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
nmol/l*min | 45.8 (7.9) | 42.6 (6.6)

4. Secondary Outcome: AUC C-peptide
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: nmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
nmol/l*min | 171.5 (16.5) | 159.2 (17.3)

5. Secondary Outcome: AUC Glucagon
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: pmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
pmol/l*min | 6933 (1056) | 7004 (1124)

6. Secondary Outcome: AUC Total GLP-1
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: pmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
pmol/l*min | 748 (115) | 1143 (218)

7. Secondary Outcome: AUC Total GIP
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: pmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
pmol/l*min | 6242 (645) | 7523 (548)

8. Secondary Outcome: AUC Active GLP-1
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: pmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
pmol/l*min | 607.9 (97.1) | 418.4 (75.6)

9. Secondary Outcome: AUC Active GIP
Time Frame: Approximately 6 weeks (range 9 - 60 days / 8.5 weeks)
Measure: Mean (Standard Error); unit: pmol/l*min
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 16 | 16
pmol/l*min | 6270 (441) | 3496 (623)

ADVERSE EVENTS:
Time Frame: up to 32 days after randomisation
Groups:
- Sitagliptin: Substance: Sitagliptin phosphate 1H2O Pharmaceutical form: tablets Source: MSD SHARP & DOHME GMBH, Doses: 100 mg, Route of administration: p.o. as a tablet
  Sitagliptin
  Mixed meal test: Subjects will be instructed to consume the mixed meal test within 20 minutes. The exact start and stop time of the mixed meal test consumption will be recorded in the CRF. The mixed meal test procedures will be identical for all subjects randomised in the study. To detect the plasma glucose excursion after mixed meal test, plasma glucose will be closely monitored
  Liraglutide: Patients on metformin monotherapy will, after screening and randomization, enter a run-in period of 2 weeks with the additional treatment of liraglutide (0.6 mg/d for 1 week followed by 1.2 mg/d for another week) that will be continued for the entire duration of the study.
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=16) | Placebo (N=16)
Headache (General disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (15) | 0 (0)
asympomatic hyppglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Results may not be interpretable for combinations of other DPP-4 Inhibitors than sitagliptin in combination with other (especially short-acting) GLP-1 receptor agonists

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No